CLINICAL TRIAL: NCT04312386
Title: Fostering Sustainable Dietary Habits Through Optimized School Meals - an Intervention Study in Uppsala, Sweden
Brief Title: Fostering Healthy and Sustainable Diets Through School Meals (OPTIMAT Uppsala)
Acronym: OPTIMAT-U
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: The Swedish Research Council for Environment, Agricultural Sciences and Spatial Planning (FORMAS) (Other Government); Göteborg University (Other)
Responsible Party: Principal Investigator, Liselotte Schäfer Elinder, professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2020-00353
Record Dates: First submitted 2020-01-21; First posted 2020-03-18 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Food Habits
Keywords: Children; Public meals; Sustainable diets; Agenda 2030; Greenhouse gas emissions
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Four schools from one county Sweden meet inclusion criteria and are eligible to participate in the intervention. These schools will all serve the baseline menu followed by the new menu. Each period will last for four weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A new 4-week lunch menu (Experimental): Optimized lunch menu with 30% lower greenhouse gas emissions, nutritionally adequate
  Interventions: Other: OPTIMAT

INTERVENTIONS:
Other: OPTIMAT — Baseline menue, not optimized

SUMMARY:
School meals have considerable potential to shape children's diets and reduce the climate impact of meals. This study applies linear programming for developing and implementing a climate friendly, nutritious and affordable school lunch menu. The new menu plan will be compared to the baseline menu during a 4-week intervention trial. The outcomes will be food waste, consumption, and pupils' satisfaction with the meals before and after introducing the new meal plan analyzed by interrupted time series analysis. Our hypothesis is that school meals can be optimized to be nutritious and more climate friendly, without negatively affecting acceptance, food waste and cost.

Four primary schools in one Swedish municipality with the same menu plan for all schools will participate in the study. Their current meal supply will be recorded in the form of a food list including amount and cost of each item over a 4-week period. This list will then be optimized with linear programming to be as similar as possible to the baseline diet but with a reduction in greenhouse gas emissions of about 30%. No new foods will be introduced and none will be removed from the list. Nutritionally adequacy will be ensured by including constraints into the model. The optimized food list will be handed to the municipality's meal planner and a new menu plan will be developed based on the revised food list. Data on food waste and consumption will be collected daily during a baseline period of four weeks, and during the four-week intervention period. School lunch satisfaction will be assessed twice with an online questionnaire at baseline and during the intervention.

DETAILED DESCRIPTION:
For a period of four weeks, during the spring term of 2020, children from four primary schools in Uppsala municipality will receive a new school lunch menu plan which has been optimized through linear programming to be as similar as possible to the baseline menu while having about 30% lower greenhouse gas emissions (GHGE), being nutritionally adequate, and not more expensive.

During the fall of 2019, a meeting was held with the public meal administration in the municipality of Uppsala. The research team described the OPTIMAT project, including the previously developed strategy for optimizing and implementing more climate friendly lunches in schools. Following this meeting, the municipality agreed to take part in the project. The municipality's meal planner proposed four primary schools for the study, presently having the highest food related GHGE in public meals in the municipality. To be eligible, the intervention schools were required to have on-site kitchens as well as being able to provide electronic recipes for a standard four-week menu. All proposed schools fulfilled these criteria and approved participation.

Recipes for an original (baseline) four-week school lunch menu plan previously served at the recruited schools were obtained through the municipality's electronic meal planning system. The foods included and amounts are considered as the baseline food supply. Each food item included has a code that can be coupled to the Swedish national food database and a national climate database for foods containing life cycle data for each food item. This baseline food supply will be optimized using linear programming. The optimized food list, not including new foods or excluding any foods from the baseline list, will be handed to the municipality's meal planner who develops a new menu plan for the intervention using all foods on the optimized list.

To assess the effect of the new menu plan, data on food waste and consumption will be collected daily in each intervention school four weeks before (baseline) as well as during the four-week intervention with a one-week brake between measurement periods. Kitchen staff will perform daily weighting (using school kitchen scales) of all food prepared in the kitchen (prepared food); the share of the prepared food that is not eaten and has to be thrown away (serving waste); the share that can be saved (leftover food); and plate waste. Total plate waste, plate waste per pupil, serving waste, total consumption, and consumption per pupil will be considered as the primary outcomes as they are regarded as directly related to the pupils' acceptability of the new menu. Data on school meal satisfaction will also be collected through an anonymous online questionnaire at baseline and during the last week of the intervention period. Pupils in grade 8 will answer the questionnaire containing ten questions related to the school lunch.

ELIGIBILITY:
Inclusion Criteria:

Primary schools (children between 6-16 years in school years 0-9)

* The schools needed to have on-site kitchens
* The schools needed to be able to provide previously used recipes for a standard four-week menu electronically

Exclusion Criteria:

Preschools or gymnasiums

* Schools receiving catered food
* Schools that could not provide recipes electronically

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2000 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in plate waste between baseline and intervention periods measured with kitchen-scales | During four weeks before the intervention period and during the four week intervention
  Plate waste, total per school and per pupil assessed with the School Food Sweden's consumption and waste measurement tool
Change in serving waste between baseline and intervention periods measured with kitchen-scales | During four weeks before the intervention period and during the four week intervention
  Serving waste, total per school assessed with the School Food Sweden's consumption and waste measurement tool
Change in food consumption between baseline and intervention periods | During four weeks before the intervention period and during the four week intervention
  Food consumption, total per school and per pupil assessed with the School Food Sweden's consumption and waste measurement tool
Change in school meal satisfaction between baseline and intervention periods | Once during the four weeks preceding the intervention as well as once during the last week of intervention
  Pupils' rating of school meals with the School Food Sweden's student questionnaire (ten questions referring to the school lunch with good face validity and with a varying number of response options from always to never or number of times per week)

SECONDARY OUTCOMES:
Change in prepared food between baseline and intervention periods measured with kitchen-scales | During four weeks before the intervention period and during the four week intervention
  Prepared food, total per school assessed with the School Food Sweden's consumption and waste measurement tool
Change in leftover food between baseline and intervention periods | During four weeks before the intervention period and during the four week intervention
  Leftover food, total per school assessed with the School Food Sweden's consumption and waste measurement tool
Change in number of lunch consumers between baseline and intervention periods | During four weeks before the intervention period and during the four week intervention
  Number of lunch consumers, total per school

CONTACTS AND LOCATIONS:
Overall Officials: Liselotte Schäfer Elinder, PhD, Principal Investigator — Karolinsk Institutet; Patricia Eustachio Colombo, MMsc., Study Chair — Karolinsk Institutet
Locations (1):
- Liselotte Schäfer Elinder, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Eustachio Colombo P, Patterson E, Schafer Elinder L, Lindroos AK, Sonesson U, Darmon N, Parlesak A. Optimizing School Food Supply: Integrating Environmental, Health, Economic, and Cultural Dimensions of Diet Sustainability with Linear Programming. Int J Environ Res Public Health. 2019 Aug 21;16(17):3019. doi: 10.3390/ijerph16173019. PMID 31438517

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-21): https://cdn.clinicaltrials.gov/large-docs/86/NCT04312386/Prot_SAP_000.pdf